CLINICAL TRIAL: NCT06990269
Title: A Phase 2, Randomized, Masked, Placebo-Controlled Study of Subcutaneously Administered ADX-038 in Participants With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: Phase 2 Study of ADX-038 in Participants With Geographic Atrophy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ADARx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-038-202
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy Secondary to Age-related Macular Degeneration
MeSH Terms: interventions — RNA, Small Interfering

STUDY DESIGN:
Intervention Model Description: Randomized, Masked, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active - ADX-038 (Experimental): Participants who meet screening eligibility criteria will be randomized to 1 of 2 treatment groups in a 2:1 ratio.
  Interventions: Drug: ADX-038
- Placebo - Saline (Placebo Comparator): Participants who meet screening eligibility criteria will be randomized to 1 of 2 treatment groups in a 2:1 ratio.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-038 — siRNA duplex oligonucleotide
  Other Names: siRNA
  Arms: Active - ADX-038
Drug: Placebo — Saline
  Arms: Placebo - Saline

SUMMARY:
Phase 2 study is designed to assess the efficacy of ADX-038 compared with placebo in participants with GA secondary to AMD. Safety, pharmacokinetics (PK), and pharmacodynamics (PD) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of GA of the macula secondary to AMD
* GA lesions between 2.5 and 12.5 mm2 at screening
* Sufficiently clear ocular media, adequate pupillary dilation and fixation to permit quality fundus imaging in the study eye as described in the protocol
* Willing and able to comply with clinic visits and study-related procedures, including completion of the full series of meningococcal vaccinations and pneumococcal vaccination required per protocol

Exclusion Criteria:

* Has GA secondary to causes other than AMD
* Has active ocular disease that compromises or confounds visual function
* History of surgery for retinal detachment
* Has ocular condition other than GA secondary to AMD
* Use of intravitreal complement inhibitors in study eye
* Hereditary or acquired complement deficiency
* Active viral, bacterial or fungal infection
* Liver injury as evidenced by abnormal liver function tests
* Donating blood
* History of choroidal neovascularization in the study eye

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of ADX-038 on the preservation of the EZ layer | 12 months
  Rate of change in the area of total EZ loss in the study eye from baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Nora Dimon, MD, Study Director — ADARx Pharmaceuticals, Inc.
Locations (17):
- United States (12):
  - ADARx Clinical Site, Gilbert, Arizona
  - ADARx Clinical Site, Phoenix, Arizona
  - ADARx Clinical Site, Beverly Hills, California
  - ADARx Clinical Site, Huntington Beach, California
  - ADARx Clinical Site, Poway, California
  - ADARx Clinical Site, Orlando, Florida
  - ADARx Clinical Site, Hagerstown, Maryland
  - ADARx Clinical Site, Erie, Pennsylvania
  - ADARx Clinical Site, McAllen, Texas
  - ADARx Clinical Site, Round Rock, Texas
  - ADARx Clinical Site, San Antonio, Texas
  - ADARx Clinical Site, The Woodlands, Texas
- Australia (3):
  - ADARx Clinical Site, Albury, New South Wales
  - ADARx Clinical Site, Parramatta, New South Wales
  - ADARx Clinical Site, Rowville, Victoria
- Canada (2):
  - ADARx Clinical Site, Ottawa, Ontario
  - ADARx Clinical Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided